CLINICAL TRIAL: NCT03112278
Title: Clinical Evaluation of Ultrathin Occlusal Veneers for the Treatment of Severe Dental Erosion
Acronym: UOVTDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Luis Henrique Schlichting, Assistant Professor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-26/112.046
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Tooth Erosion; Teeth Erosion Due to Vomiting; Teeth Erosion Limited to the Enamel; Teeth Erosion Extending Into the Dentine
Keywords: tooth erosion; Computer-Aided Design; occlusal veneers; dental veneers
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both patient and the evaluators that will asses the performance of the restorations are unaware about the type of material used to fabricate the occlusal veneers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceramic restorations (Active Comparator): Ceramic ultrathin occlusal veneers
  Interventions: Procedure: Ceramic ultrathin occlusal veneers
- Composite resin restorations (Active Comparator): Composite resin ultrathin occlusal veneers
  Interventions: Procedure: Composite resin ultrathin occlusal veneers

INTERVENTIONS:
Procedure: Ceramic ultrathin occlusal veneers — Severely eroded teeth will be restored with ultrathin occlusal veneers made of ceramic (e.max CAD/Ivoclar Vivadent) by technology CAD-CAM bonded to the teeth (0.6 - 1.2 mm thick).
  Arms: Ceramic restorations
Procedure: Composite resin ultrathin occlusal veneers — Severely eroded teeth will be restored ultrathin occlusal veneers made of composite resin (Lava Ultimate/3M Espe) by technology CAD-CAM bonded to the teeth (0.6 - 1.2 mm thick).
  Arms: Composite resin restorations

SUMMARY:
Ultra-thin bonded posterior occlusal veneers represent a conservative alternative to traditional onlays and complete coverage crowns for the treatment of severe erosive lesions. Therefore, the purpose of this study is to determine whether ceramic and composite resin ultrathin occlusal veneers (0.6 - 1.0 mm thick) are effective in the rehabilitation of patients affected by moderate and severe dental erosion.

DETAILED DESCRIPTION:
Along with data collection, complete arch polyvinyl siloxane impressions are made to obtain accurate diagnostic casts. The occlusal relationship is recorded either at the maximum intercuspal position or centric relation (in cases occlusal space is needed for the restoration of the palatal of upper anterior teeth). An additive waxing is carried out for the eroded teeth. The waxed cast is then duplicated and poured with scannable stone.

An average occlusal clearance of 0.4 to 0.6 mm (central groove) to 1.0 to 1.3 mm (cusp tips) is generated by means of rotary diamond burs for the ultrathin occlusal veneers. A rubber dam is placed, and all areas of dentin exposure are ground with a coarse diamond rotary instrument at low speed (1500 rpm) and immediately sealed using a 3-step etch-and-rinse dentin bonding agent. The additive wax replica is scanned first for correlation (Cerec Bluecam; Sirona Dental Systems). The prepared teeth are then scanned in the same way.

The teeth are restored using Cerec AC with the Bluecam/MCXL CAD/CAM system (Sirona Dental Systems). By using the design tools of the software set in Biogeneric Copy, the restorations are designed by correlating the preparations with the anatomy of the additive waxing. The ultrathin occlusal veneers are milled either from composite resin blocks (LAVA Ultimate; 3M ESPE) or ceramic blocks (e.max CAD; Ivoclar Vivadent) and polished mechanically with silicon carbide-impregnated brushes.

Restorations are then adhesively cemented. After being air-dried, the intaglio surfaces are silanated and heat dried at 68 oC for 5 minutes (Calset; AdDent Inc). The tooth preparations are airborne-particle abraded and etched for 30 seconds with 37.5% phosphoric acid, rinsed, and dried. Adhesive resin (Optibond FL, bottle 2; Kerr Corp) is applied to both fitting surfaces of the restoration. After the luting material (Filtek Z100; 3M ESPE), preheated to 68oC (in Calset; AdDent), is applied to the tooth, the restorations were individually seated, followed by the elimination of excess composite resin and initial light polymerization. Each surface is exposed at 1000 mW/cm2 for 1 minute (20 seconds per surface, repeated 3 times). Margins are then covered with an air barrier and light polymerized for an additional 20 seconds. Margins are finished and polished at the following appointment with diamond ceramic polishers and silicon impregnated rubber polishers.

Patients are called for a base line evaluation followed by additional evaluations after 1 year, 2 years and 4 years.

Patients Registries:

Patients' registries are made in paper forms and immediately digitalized for safety. The form is stored inside an identified folder containing other patient's documents related to the treatment.

Upon completion of the registry all data is verified by a third person to check for completeness, calibration and accuracy.

Two researchers linked to the project perform patient recruitment (not the evaluators). Patients are interviewed and seen for data collection. If eligibility criteria are meet, the patient receives a comprehensive explanation (accessible language) about the protocol and an invitation to participate.

Despite evaluators were previously calibrated; detailed description of the criteria (based on USPHS) is available to the evaluator at every data collection (follow-up appointments).

Patients are seen at clinic of the Department of Prosthodontics and Dental Materials of the Dental School of UFRJ. During the follow-up appointments data is collected in sequence by two calibrated evaluators. In case of divergence, a consensus is achieved. Intraoral evaluation is performed with dental explorer and mouth mirror assisted by dental operatory light as well as well as a LED transilluminator for crack chasing. In case of failure (cracks longer than 2 mm, lost fragments or bulk debondings) patients are assigned for repair or change of restoration.

The sample of 5 patients for each group was based on the following formula: n = (Zα/2+Zβ)2 * (p1(1-p1)+p2(1-p2)) / (p1-p2)2, with a confidence level of 95%, power of 80% and the survival rates of 90% and 20% for composite and ceramic restorations, respectively (based on previous published data of in vitro fatigue tests).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting advanced erosive lesions ( cumulative score in all sextants greater than or equal 14, according to classification of BARLETT; GANSS; LUSSI, 2008).
* Absence of pain from the tooth to be restored (excluding expected sensitivity due to dentin exposure due to severe erosion).
* Application of rubber dam possible
* High level of oral hygiene.
* Absence of any active periodontal and pulpal disease.
* Willingness to wear a nightguard to protect the restorations in case of associated bruxism.

Exclusion Criteria:

* patients with low level of oral hygiene after all the attempts to improve it failed.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2021-04-02 (Estimated)

PRIMARY OUTCOMES:
Survival of ultrathin occlusal veneers (ceramic and composite resin) for the restorative treatment of severe dental erosion. | 1Year

CONTACTS AND LOCATIONS:
Overall Officials: Luis H Schlichting, PhD, Principal Investigator — Federal University of Rio de Janeiro and East Carolina University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bindl A, Mormann WH. Survival rate of mono-ceramic and ceramic-core CAD/CAM-generated anterior crowns over 2-5 years. Eur J Oral Sci. 2004 Apr;112(2):197-204. doi: 10.1111/j.1600-0722.2004.00119.x. PMID 15056119
- [Background] Burke FJ. Maximising the fracture resistance of dentine-bonded all-ceramic crowns. J Dent. 1999 Mar;27(3):169-73. doi: 10.1016/s0300-5712(98)00050-5. PMID 10079622
- [Background] Edelhoff D, Sorensen JA. Tooth structure removal associated with various preparation designs for posterior teeth. Int J Periodontics Restorative Dent. 2002 Jun;22(3):241-9. PMID 12186346
- [Background] Edelhoff D, Sorensen JA. Tooth structure removal associated with various preparation designs for anterior teeth. J Prosthet Dent. 2002 May;87(5):503-9. doi: 10.1067/mpr.2002.124094. PMID 12070513
- [Background] Fennis WM, Kuijs RH, Kreulen CM, Verdonschot N, Creugers NH. Fatigue resistance of teeth restored with cuspal-coverage composite restorations. Int J Prosthodont. 2004 May-Jun;17(3):313-7. PMID 15237878
- [Background] Jaeggi T, Lussi A. Prevalence, incidence and distribution of erosion. Monogr Oral Sci. 2006;20:44-65. doi: 10.1159/000093350. PMID 16687884
- [Background] Kunzelmann KH, Jelen B, Mehl A, Hickel R. Wear evaluation of MZ100 compared to ceramic CAD/CAM materials. Int J Comput Dent. 2001 Jul;4(3):171-84. English, German. PMID 11862884
- [Background] Leinfelder KF. Ask the expert. Will ceramic restorations be challenged in the future? J Am Dent Assoc. 2001 Jan;132(1):46-7. doi: 10.14219/jada.archive.2001.0024. No abstract available. PMID 11194398
- [Background] Lussi A, Hellwig E, Ganss C, Jaeggi T. Buonocore Memorial Lecture. Dental erosion. Oper Dent. 2009 May-Jun;34(3):251-62. doi: 10.2341/09-BL. PMID 19544813
- [Background] Magne P. Composite resins and bonded porcelain: the postamalgam era? J Calif Dent Assoc. 2006 Feb;34(2):135-47. PMID 16724469
- [Background] Magne P, Schlichting LH, Maia HP, Baratieri LN. In vitro fatigue resistance of CAD/CAM composite resin and ceramic posterior occlusal veneers. J Prosthet Dent. 2010 Sep;104(3):149-57. doi: 10.1016/S0022-3913(10)60111-4. PMID 20813228
- [Background] Manhart J, Chen H, Hamm G, Hickel R. Buonocore Memorial Lecture. Review of the clinical survival of direct and indirect restorations in posterior teeth of the permanent dentition. Oper Dent. 2004 Sep-Oct;29(5):481-508. PMID 15470871
- [Background] Magne P, Stanley K, Schlichting LH. Modeling of ultrathin occlusal veneers. Dent Mater. 2012 Jul;28(7):777-82. doi: 10.1016/j.dental.2012.04.002. Epub 2012 May 9. PMID 22575740
- [Background] Schlichting LH, Maia HP, Baratieri LN, Magne P. Novel-design ultra-thin CAD/CAM composite resin and ceramic occlusal veneers for the treatment of severe dental erosion. J Prosthet Dent. 2011 Apr;105(4):217-26. doi: 10.1016/S0022-3913(11)60035-8. PMID 21458646
- [Background] Tsitrou EA, van Noort R. Minimal preparation designs for single posterior indirect prostheses with the use of the Cerec system. Int J Comput Dent. 2008;11(3-4):227-40. English, German. PMID 19216314
- [Background] Vailati F, Belser UC. Full-mouth adhesive rehabilitation of a severely eroded dentition: the three-step technique. Part 1. Eur J Esthet Dent. 2008 Spring;3(1):30-44. PMID 19655557
- [Result] Schlichting LH, Resende TH, Reis KR, Magne P. Simplified treatment of severe dental erosion with ultrathin CAD-CAM composite occlusal veneers and anterior bilaminar veneers. J Prosthet Dent. 2016 Oct;116(4):474-482. doi: 10.1016/j.prosdent.2016.02.013. Epub 2016 Apr 29. PMID 27132785